CLINICAL TRIAL: NCT03428464
Title: Bicarbonate Administration in Kidney Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17-2317
Record Dates: First submitted 2018-01-29; First posted 2018-02-09 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Kidney Transplant; Complications; Metabolic Acidosis
MeSH Terms: conditions — Acidosis | interventions — Sodium Bicarbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sodium bicarbonate (Experimental): During the treatment period, participants will receive 0.5 mEq/kg-lean body weight (LBW)/day of oral sodium bicarbonate for 8 weeks.
  Interventions: Drug: Sodium Bicarbonate
- Placebo (Placebo Comparator): During the control period, participants will take the same number of placebo capsules as if they were assigned 0.5 mEq/kg-LBW/day of sodium bicarbonate.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Sodium Bicarbonate — Participants will take ½ the daily dose of sodium bicarbonate in the morning and the other ½ in the evening.
  Other Names: Baking soda
  Arms: Sodium bicarbonate
Other: Placebo — Participants will take ½ the daily dose of a placebo in the morning and the other ½ in the evening.
  Arms: Placebo

SUMMARY:
Metabolic acidosis is associated with vascular endothelial dysfunction and is a common complication in patients who have received a kidney transplant. Kidney transplant recipients (KTR) with lower serum bicarbonate levels, even within the normal range, have an increased risk of graft loss and mortality. The investigators propose a prospective, double-blind, randomized, placebo-controlled, 18-week crossover pilot study to examine the effects of sodium bicarbonate on vascular endothelial function, graft function, and cognitive function in 20 KTR patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Kidney transplant received at least 1 year ago
* Serum bicarbonate 20-26 mEq/L on 2 separate measurements (at least 1 day apart)
* eGFR >45 ml/min/1.73m2
* Blood pressure <140/90 mm Hg prior to randomization
* BMI < 40 kg/m2 (FMD measurements can be inaccurate in severely obese patients).
* Able to provide consent
* Stable kidney transplant medication regimen for at least 1 month prior to randomization
* Stable anti-hypertensive regimen for at least one month prior to randomization
* Not taking medications that interact with agents administered during experimental sessions (e.g. sildenafil interacts with nitroglycerin).

Exclusion Criteria:

* Significant comorbid conditions that lead the investigator to conclude that life expectancy is less than 1 year
* Use of chronic daily oral alkali within the last 3 months (including sodium bicarbonate, calcium carbonate or baking soda)
* Uncontrolled hypertension
* Serum potassium < 3.3 or ≥ 5.5 mEq/L at screening
* New York Heart Association Class 3 or 4 heart failure symptoms, known EF ≤30%, or hospital admission for heart failure within the past 3 months · Factors judged to limit adherence to interventions
* Current participation in another research study
* Pregnancy or planning to become pregnant or currently breastfeeding
* Chronic use of supplemental oxygen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2020-03-25 (Actual)

PRIMARY OUTCOMES:
Change in Brachial Artery Flow-Mediated Dilation | Baseline, 8, 10, and 18 weeks
  Brachial artery Flow-Mediated Dilation (FMD) will be determined using high-resolution ultrasonography (Toshiba Xario 200) as described originally by Celermajer et al., and more recently by our group. FMD will be measured at the beginning and end of each study period for a total of 4 measurements. ECG-gated end-diastolic ultrasound images and Doppler flow of the brachial artery will be acquired during baseline and FMD conditions.

SECONDARY OUTCOMES:
Change in Transforming Growth Factor Beta 1 (TGF-B1) | Baseline, 8, 10, and 18 weeks
  Urinary TGF-B1 will be measured from 24-hour urine collections. It will be measured by a commercially available ELISA (R&D Systems). The within day precision for this assay is 6.7% at 257 pg/ml. All measurements will be performed at the Children's Pediatric CTRC at Children's Hospital Colorado.
Change in Cognitive Function | Baseline, 8, 10, and 18 weeks
  Cognitive function will be assessed using the National Institutes of Health (NIH) Toolbox computerized tests to evaluate 1) attention, 2) episodic memory, 3) working memory, 4) language, 5) executive function, and 6) processing speed.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Kendrick, MD MPH, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States